CLINICAL TRIAL: NCT04169334
Title: A Family Focused and Optimized Postpartum Programme at the Obstetric Department and Across Sectors for Vulnerable Families. - A Mixed-method Study of the Obstetric Care Delivered to Vulnerable Families in Order to Foster an Early Healthy Relationship Formation.
Brief Title: Look - Your Baby is Talking to You.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Camilla Ejlertsen, PhD student, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-18021300
Record Dates: First submitted 2019-11-11; First posted 2019-11-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Intervention study with one controlgroup and one intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Group receiving care as usual
- Intervention group (Experimental): Intervention group receiving a standardized preventive program (5 days at the Obstetric department)
  Interventions: Behavioral: Prolonged planned program for the stay at the obstetric department

INTERVENTIONS:
Behavioral: Prolonged planned program for the stay at the obstetric department — A five day planned and designed program delivered to the family while at the obstetric department.
  Arms: Intervention group

SUMMARY:
It is well documented that the formation of the early relation between parents and infant has a significant impact on the child's mental, social and cognitive development and competencies. The early relationship formation in the first year in the infants' life gets the best conditions when parents are able to interpret, understand and respond to the infants signal adequately. Symptoms of mental illness can affect a person's ability to respond to their environment and thereby their parenting capabilities. Research have found that parental psychopathology may interfere with a healthy interaction with the infant by reducing the ability to be sensitively attuned and responsive to the infant's signal, needs and cues due to the nature of the psychiatric symptoms.

The aim of this study is to investigate what potential lies within the postpartum stay at the obstetric department and in the transition to the primary health care sector for vulnerable families and to develop an intervention that will help increase the parents sensitivity towards their new born infant in order to enter a healthy early relationship formation which will be measureable on short term in the prevalence of maternal post-partum depression.

The study is a prospective mixed-method study consisting of three sub-studies. The first study is a register-based study which aims to investigate how the proportion and the absolute risk of children with predefined adverse developmental outcomes is distributed between families defined as level three or four compared to families defined as level one and two. The second study aims to uncover needs and preferences of the vulnerable families and to investigate the experiences of the health care professionals. It is explored by in-depth family interviews with families discharged from the obstetric department and focus group interviews with health care professionals (nurses and health visitors) who are responsible for the care delivered to vulnerable families. Subsequently an intervention study will be developed, adapted, implemented and evaluated. The intervention will be carried out at the obstetric department at Hvidovre hospital and in transition to the primary healthcare sector using components from family focused nursing (FFN) and neonatal behavioral observational sessions (NBO) in addition to what have appeared in the two first sub-studies. The aim of the intervention is to facilitate family consciousness of their resources'' and increase parental sensitivity in order to foster the best possible prerequisites for a healthy early relationship formation between parent and infant.

The study population consists of mothers with anxiety or depression diagnosis giving birth at Hvidovre hospital.

The register-based study will provide population based information on the characteristics of vulnerable families focusing on the adverse outcomes for the children. The qualitative interviews will contribute with in-depth knowledge about preferences and experiences in relation to the care offered within the extended stay at the obstetric department and in the transition to primary health care sector and everyday life for vulnerable families.

The enactment, implementation and evaluation of the intervention will determine whether the combination of FFN, NBO and improved collaboration between the obstetric department and the health visitor is associated with increased family function and increased parental sensitivity among parents in the intervention group compared to the control group. Effect from baseline (24-48 hours post-partum) to follow-up (3 months post-partum) will be measured on both the mother, the parents and the infant focusing on depression symptoms (primary outcome), parental stress, parental reflective function, mother-baby interaction, couple relationship satisfaction, infants' self-regulation, family function and breastfeeding Descriptive statistics will be applied in order to detect associations. Power calculations showed that with a significance level of 5% and a power of 80% 55 families are needed in the control and the intervention group, respectively, in order to detect statistically difference.

This PhD study will contribute with a new perspective on the potential of the time immediately after birth and the potential effect of early intervention to improve prerequisites for increased family function and early healthy relationship formation for vulnerable families. The study will provide knowledge and experience about the practical application of both FFN and NBO at the obstetric department which have never been done in a Danish context before. It is expected that the study as a whole may impact and benefit clinical nursing as well a public health.

DETAILED DESCRIPTION:
Background The formation of the early relation between parents and infant has a significant impact on the infant's mental, social and cognitive development and competencies. Parental psychopathology may interfere with a healthy interaction by reducing the ability to be sensitively attuned to the infant's signal and needs due to the nature of the psychiatric symptoms. A healthy psycho-social development starts in the perinatal period in which the parent-infant interactions comprise of one of the most influential experiences which make infants vulnerable and exposed to mental health risks in a lifespan perspective. International research has found that the consequences of being born by a mother suffering from mental illness influences on the infant's risks of developing psychopathology, developmental disorders, and problems related to the social negative heritage. In order to initiate preventive programs, the long-term effects of being born by a vulnerable mother need to be investigated to target and design effective interventions. In a Danish context it is also of interest to investigate how the proportions of children with poorer developmental outcomes are distributed between vulnerable and not-vulnerable families.

It is well-documented that early intervention improves the prognosis for infants of vulnerable families and short-term programs consisting of a moderate number of sessions aimed at improving interaction are especially effective in enhancing parental sensitivity and infant attachment security. Furthermore, the World Health Organization recommends that new families are supported in the development of a healthy parent-infant relationship. The postpartum period has been identified as particularly important for the establishment of early healthy parent-infant relationship and health professionals at the obstetric department (obs. dept.) and health visitors in the primary health care sector are in a perfect position to initiate intervention programs that enhances this. Understanding and identifying the quality of the parent-infant relationship is important in both hospital setting and in the primary health care sector which also demands knowledge-sharing across sectors to create coherence. In Denmark the antenatal care is differentiated according to the recommendations from the National Board of Health, offering families categorized as level three and four an extended stay at the obs. dept. following birth. Level three covers vulnerable families comprising of families experiencing social, medical or psychological problems such as e.g. anxiety or depression. Level four covers families experiencing complicated and severe problems with drug abuse or severe psychiatric disorders. These families are offered an extended stay at the obs. dept. which in most Danish hospitals are 5 days.

It is estimated that around 10-14 percentage (n= 980) of families giving birth at Hvidovre Hospital (HVH) are vulnerable. The care and the content of the extended stay is based on recommendations, and is not standardized. Further it has not been investigated what the families' preferences and wishes for the extended stay consists of or what the health professionals experience when taking care of vulnerable families at the obs. dept. The transition to the primary health care sector is also not standardized and trading of information and observation are not ensured.

Vulnerable families need support in the relationship formation . A mentally ill mother demands activation and involvement of the family as a resource to facilitate the best possible prerequisites for a healthy relationship formation with the infant. Substantial evidence have formed an understanding that treatment of postnatal depression might require specific parenting components to benefit child outcome. In addition, some studies have found that intervention programs designed specifically towards improvement of the mother-infant relationship in the context of postnatal depression benefit both the relationship formation and reduces the negative effects of maternal depression on child development. Therefore it is assumed that a combination of a family approach assessing family resources and a relationship based tool that helps parents read their infants self-regulatory cues resulting in an enhanced relationship-formation may decrease the prevalence of maternal post-partum depression.

Aim The aim of this study is to investigate how the extended postpartum stay at the obs. dept. and the transition to the primary health care sector can be optimized for vulnerable families. Furthermore, to develop and test an intervention program that aim to increase parental sensitivity and facilitate a healthy early relationship formation with their infant which may reduce depressive symptoms among vulnerable mothers.

The aim of the study will be achieved by answering the following research questions:

1. To which extent can adverse child developmental outcomes be predicted by the vulnerability groups?
2. How do health care professionals experience the extended stay at the obstetric department and the transition to the primary healthcare sector?
3. Does a standardized program offered at the obstetric department containing elements from NBO and FFN and a systematic transition to primary health care improve prerequisites for a healthy early relationship formation between parents and infant and thereby reduced depressive symptoms among vulnerable mothers?

Sub-study 1: Register-based study Being born by a vulnerable mother is associated with adverse child developmental outcomes and being born into a vulnerable family may have wide ranging effects on child development. These effects include impairment in cognitive performance, behavior disturbances and mental problems that may persist into late childhood and adolescence. However, it is of interest to investigate if the classification of vulnerable groups, the strategy used by the antenatal care to predict vulnerable groups and designing intervention programs only aiming at these groups is enough.

This study aim to investigate how the proportion and the absolute risk of children with predefined adverse developmental outcomes is distributed between families defined as level three or four compared to families defined as level one and two according to the to the antenatal care defined by The National Board of Health . Adverse child developmental outcomes will be defined completion of ninth grade before age 18, grade point average at the ninth-grade exams in Danish public and private schools and social professional interventions in the home. The study is conducted as a national register-based cohort study with a study population consisting of all Danish children born from 1980-2015. Data will be extracted from the Medical Birth Registry, the Danish National Patient Registry and Statistics Denmark's Registries. Descriptive statistics will be applied using STATA (StataCorp. 2015). The study will be carried out in collaboration with an epidemiological research unit at the University of Copenhagen that has great experience with register-based research.

Sub-study 2: Interviews The interview-study aim to uncover the experiences of the health care professionals.

Focus group interviews. Two focus group interviews (FGI) will be held of 2 hours respectively. Both with 3-5 nurses from the obs. dept. and 3-5 health visitors from collaborating municipalities. In total 12-20 participators.

The FGI will take place at the hospital and will be facilitated by two researchers (PhD student and senior researcher). An interview-guide will be developed to guide the discussions and the FGI will be digitally recorded. Data will be analyzed using content analysis

Sub-study 3: Intervention study The intervention study is designed as a feasibility study, that aim to test and put the developed intervention program into practice. The study will investigate enquiries related to content, recruitment, applicability of the outcome measures, time-frame and follow-up period, reasoning and adaptability of statistics. Further the study is unique in terms of complexity and collaboration across sectors. The health professionals from the obs. dept. will be trained to carry out the intervention program. Data on the on the control group will be collected prior launch of the intervention program to prevent bias and to ease the logistic concerning organization of the health professionals at the obs. Dep. The control group consists of women giving birth at HVH meeting the same criteria as the intervention group and they will receive care as usual.

The intervention program comprises of results and knowledge gathered from sub-study 1 and 2, standardized transition to primary health care sector and the beneath listed components:

Family-focused nursing. The theoretical framework is the philosophy of Family Centered Care (FCC). It embraces respect and equality, shared responsibility, knowledge-sharing, cooperation and partnership between health care professionals and families. Family Focused nursing (FFN) is the practical application of delivering FCC. Assessing family resources, coping strategies and processes relating to relations and communications among family members, through FFN conversations provides the foundation of assisting families in their adaption and attainment of a higher level of family function, support, health and well-being. FFN conversations are based on systems theory, change theory and communication theory using genograms to map the structure of the family and used as a basis for the subsequent interventions.

Newborn behavioral observation System (NBO) The NBO is an individualized, infant-focused, family-centered and systematic observational system that is designed to be used by health professionals to assist, elicit and describe the newborns' competencies and individuality, with the explicit goal of strengthening the relationship between parents and the infant and it has been developed as a means of supporting parents in the transition to parenthood. The NBO system comprises of 18 neuro-behavioral observations of the infant when sleeping, being awake or crying. Combining FFN and NBO in an intervention program will increase focus on the family's resources and ensure that the infant gets an explicit voice that is thought to increase parental sensitivity and thereby decrease the risk of maternal post-partum depression.

The intervention program is thought as preventive and aim to increase parental sensitivity expressed as a lower prevalence of maternal postpartum depression symptoms. In total10 health professionals from the obs. dept. will be theoretically and practically educated in the methods: FFN (3days) and certified in the NBO (3days). The intervention program delivered to the intervention group participators consists of FFN conversations and NBO sessions that will be structured throughout the stay at the obs. dept. At the first day following birth an admission dialogue is held with the family that implies a FFN conversation. On the second, third and fourth day of the stay NBO sessions will be held with the family. On the third day the NBO session will be combined with another FFN conversation and on the last day of the stay a transition dialogue will be held together with a health visitor from the family's home municipality. This transition dialogue will contain a FFN conversation. The conversations and sessions will vary in length (but are estimated to last around 45 minutes per conversation) and content and will be shaped by the needs and preferences of the family. The transition-dialogue on the day of discharge will be held to ensure that important observations, knowledge and concerns are shared with the family and between the health professionals. Contact and formal agreements with the collaborating communities will be made prior launch of the intervention program.

Descriptive statistics will be applied using STATA (StataCorp. 2015) and T-tests, Chi2 and regression analysis will be performed and when relevant comparison will be controlled for confounding. Process evaluation is applied to ensure that the intervention program is delivered according to the intention. During the intervention period documentation for held FFN conversations and NBO sessions will be collected and ongoing evaluation will register drop-outs or recruiting problems. Besides the PhD student will randomly witness both FFN conversations and NBO sessions in order to ensure intended content.

The sample size is calculated on the basis of the difference between the control and the intervention group on the maternal Edinburg Postnatal Depression scale (EPDS) at follow-up. It is estimated that the prevalence of an elevated EPDS score will be 50% in the study population due to the inclusion criteria (42,43) and a power calculation shows that with a significance level of 5 % and a power of 80% 55 participating and followed-up families in both the control and the intervention group is needed to detect significant difference (N = 110). Ethics: Participating families are informed about the purpose of the study and will receive both oral and written information about the study prior participation. The study will be reported to the Committee on Health Research Ethics and the Danish Data Protection Agency.

Perspectives Combining research from three sub-studies this PhD study will increase the understanding of how the time immediate after birth may facilitate family consciousness of their resources' and help evolve early healthy relationship formation. This study will be the first to implement and adapt FFN and NBO to a high-risk population at an obs. dept. in Denmark. Furthermore, it is expected that this study will impact and profile clinical

ELIGIBILITY:
Inclusion Criteria:

* Mothers with ongoing or former either depression or anxiety diagnosis

Exclusion Criteria:

* Other psychiatric comorbidities
* Premature birth (<37 week)
* admission to neonatal unit
* if the infant is born with syndromes or other malformations.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women delivering at Hvidovre hospital meeting inclusion criteria
Enrollment: 121 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Change in maternal depressive symptoms from baseline to three month postpartum | Baseline and 3 month post partum
  Edinburgh postnatal depression score, rates on a four point scale from 'most of the time' to 'never' Cut off at 11. The higher the score the more depressive symptoms.

SECONDARY OUTCOMES:
Parental Stress scale | Baseline and 3 month post partum
  Measures parental stress, 18 items, The item statements are rated for agreement by parents using a 5-point response scale (1 = strongly disagree, 2 = disagree, 3 = undecided, 4 = agree, 5 = strongly agree)
Parental reflective function | Baseline and 3 month post partum
  Parental Reflective Functioning Questionnaire, 18 items, rates on a visual scale from strongly disagree to strongly agree
Family function | Baseline and 3 month post partum
  The Iceland-Expressive Family Functioning Questionnaire, 17 items, rates on a five point cale from almost never to almost always
Infant self-regulations | Baseline and 3 month post partum
  Questions regarding infant selfregulation, rates on a four point scale from never to always
Process evaluation | When the family is discharged.
  Measures if the intervention is delivered

CONTACTS AND LOCATIONS:
Locations (1):
- COpenhagen University Hospital Hvidovre, Hvidovre, Danmark, Denmark